CLINICAL TRIAL: NCT07225231
Title: Byteflies Real-world Data Study: Assessing the Clinical Utility of Reduced EEG Montage Home Monitoring for Clinician-driven Fenfluramine Titration in Dravet Syndrome and Lennox-Gastaut Syndrome
Brief Title: Clinical Utility of Reduced EEG Home Monitoring in Fenfluramine Titration for Dravet and LGS
Acronym: TETRIS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Byteflies (Industry)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BF0003
Record Dates: First submitted 2025-10-31; First posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Dravet Syndrome (DS); Lennox Gastaut Syndrome (LGS)
MeSH Terms: conditions — Epilepsies, Myoclonic; Lennox Gastaut Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Patient treated with standard-of-care fenfluramine and wearing remote patient monitoring solution (Experimental): Participants will receive standard-of-care fenfluramine treatment as prescribed for their clinical condition. In addition, they will be equipped with a remote patient monitoring (RPM) solution designed to collect EEG, ECG and EMG data.
  Interventions: Device: Byteflies Remote patient monitoring solution (with reduced EEG)

INTERVENTIONS:
Device: Byteflies Remote patient monitoring solution (with reduced EEG) — Remote patient monitoring (RPM) solution designed to collect EEG, ECG and EMG data.

SUMMARY:
The goal of this real world data study is to evaluate the clinical utility of remote patient monitoring solution (using Byteflies' EpiCare@Home with reduced EEG montage and other vital signs) with Dravet and LGS patients (ages 3 and up with the exclusion of adults above weight allowing variable titration) to identify an optimal Fenfluramine treatment.

Patients will wear one or more small portable and medically certified measuring devices. Through these devices, electroencephalography (EEG) signals, as well as electro-cardiography (ECG), heart rate, respiration rate, and physical activity are measured, which allows the patient's physician to detect potential seizures, and thus gain more insights.

Participants will be asked to wear the devices three times at home for remote monitoring periods lasting between 3 and 7 consecutive days. The duration of each monitoring period will be determined by the physician based on the type of epilepsy and the frequency of seizures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed Dravet syndrome or Lennox-Gastaut syndrome diagnosis who are eligible for Fenfluramine.
* Patients for which the neurologist decided to prescribe Fenfluramine as a relevant treatment approach and who have not been prescribed Fenfluramine before.
* Patients or caregivers should be able and willing to maintain a seizure diary e.g. using a digital seizure diary.

Exclusion Criteria: Patients who

* Have been diagnosed with or are suspected to have life-threatening conditions that could result in immediate danger;
* Need to undergo an MRI scan or cardiac defibrillation;
* Have an active implanted device such as a pacemaker, defibrillator, or vagal nerve, or brain stimulator;
* Are unable to provide written informed consent, either directly or via a legal guardian.
* Have known allergy or skin-sensitivity to the materials used in the Byteflies Adhesives
* Are between 0 and 3 years of age;
* Are above weight allowing variable titration
* The patient is on any medication that would be contra-indicated for use with Fenfluramine at the execution of the study eg. LP352 (bexicaserin), loracaserin, monoamine-oxidase inhibitors, SSRIs, SNRIs, tricyclic antidepressants or other serotonergic agonists or antagonists (antipsychotics).
* Have a prescribed concomitant use of Stiripentol
* Have any other condition or finding that would compromise the safety of the participant or the quality of the data, or otherwise interfere with achieving the objectives.
* A history of cardiovascular or cerebrovascular disease, aortic or mitral valve regurgitation diagnosed by echography
* Patients/caregivers who have only reported/detected non-motor seizures

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Physician confidence in treatment decision-making using RPM data | At end of first RPM period (2 weeks after treatment start), at end of second RPM period (between 1 to 3 months after treatment start), at end of third RPM period (between 3 to 9 months after treatment start)
  The primary endpoint of the study is defined as the proportion of cases in which physicians report higher confidence in treatment decision-making when using RPM-enhanced data compared to standard care, with increased confidence defined as an RPM confidence score greater than the standard confidence score. The primary endpoint is considered successful if physicians demonstrate improved confidence in their treatment decisions for at least 50% of the patients when RPM data is available.
  For each patient, the following assessments will be performed:
  1. Standard Decision (-RPM): Clinicians will determine the treatment plan based on routine data. Clinicians will record their confidence in this decision on a 1-5 Likert scale (1 = not confident, 5 = very confident).
  2. RPM-Enhanced Decision (+RPM): Clinicians will determine the treatment plan using the same routine data plus information provided by the RPM system. Clinicians will record their confidence in this decision on a 1-5 Likert scale.

IPD SHARING:
Plan to Share IPD: No